CLINICAL TRIAL: NCT04452409
Title: Enhanced Liver Function in Non-alcoholic Obese Fatty Liver Patients by Low Level Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ebtesam Nabil, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/002722
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Fatty Liver, Nonalcoholic; Liver Function
Keywords: low level laser
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Low-Level Light Therapy; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (low level laser plus Mediterranean diet) (Active Comparator): Active infra -red laser in addition to diet
  Interventions: Device: low level laser; Other: Mediterranean diet
- control (Mediterranean diet only) (Other): diet
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Device: low level laser — The laser therapy device (660 nm) consisted of abdominal straps containing 4 LED clusters, having 72 LEDs each, applied in the study group paticipants around the patients abdomen and waist after cleaning the target area and wearing safety goggles20, for 30 min., 2 times per week over 12 weeks
  Arms: study (low level laser plus Mediterranean diet)
Other: Mediterranean diet — recommend healthy diet component evaluated periodically by 24 hour recall

SUMMARY:
Non-alcoholic fatty liver disease is excessive fat build-up in the liver with insulin resistance due to causes other than alcohol use.The obesity epidemic is closely associated with the rising prevalence and severity of nonalcoholic fatty liver disease.Currently, the only treatment modality for patients with fatty liver disease is weight loss and exercise which is challenging for most patients. Therefore, a huge need exists for an alternative approach to reducing alanine transaminase (ALT) & aspartate aminotransferase (AST) levels for these patients. Low level laser light therapy (LLLT) offers a simple, non-invasive, safe, effective and side-effect free alternative to achieving this goal, through LLLT's proven ability to effect weight loss, body circumference reduction and lipid profile modification

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a very common disorder and refers to a group of conditions where there is accumulation of excess fat in the liver of people who drink little or no alcohol. The most common form of NAFLD is a non serious condition called fatty liver.

NAFLD is part of the metabolic syndrome characterized by diabetes, or pre-diabetes (insulin resistance), being overweight or obese, elevated blood lipids such as cholesterol and triglycerides, as well as high blood pressure. A few studies have suggested that weight loss may be associated with regression of fat within the liver. Therefore, the most important recommendations for people with fatty liver are to lose weight if they are overweight or obese, increase their physical activity, follow a balanced diet and unnecessary medications.

Several studies have investigated low-level laser therapy (LLLT) or light-emitting diode (LED) therapy and have made advances in the understanding of the underlying mechanisms LLLT in biological systems. Few studies explain the effect of low level laser therapy on liver enzymes and non alcoholic fatty liver risk factors (as obesity).So, our goal was to perform a randomized controlled trial to investigate the effects of the LLLT on lipid profile, body weight and liver enzymes

ELIGIBILITY:
Inclusion Criteria:

* • Sixty non-alcoholic fatty liver patients aged from 60-75 y

  * Body mass index (BMI) ranged from 30 to 34.9 kg/m2
  * Elevated triglyceride & LDL levels
  * Higher Risk Waist Circumference Measurements (Men: 40 or more inches or 102 centimeters or more/ Women: 35 or more inches or 89 centimeters or more)
  * Elevated aminoalanine transaminase (ALT) level, defined as 20 or more Unites/Liter (U/L) above the normal gender-specific ALT levels: males: ALT ≥ 60 U/L; females: ALT ≥ 50 U/L
  * Review of subject's pre-existing medical records to confirm the current diagnosis of nonalcoholic fatty liver according to the following criteria:
  * ALT elevated on two separate determinations
  * Abdominal ultrasound showing fatty liver
  * Blood work that excludes other potential etiologies of liver disease
  * Subject agrees to maintain his or her diet regimen throughout study participation

Exclusion Criteria:

* • History of cardiovascular disease or events including, but not limited to, coronary artery disease, valvular heart disease, cardiac arrhythmias, congestive heart failure, myocardial infarction, stroke, transient ischemic attack, or peripheral vascular disease

  * Cardiac surgeries or procedures, including but not limited to, coronary artery bypass surgery or stent placement, heart transplantation, pacemaker insertion or implantation of a defibrillator
  * An implanted device in the target area to receive low level laser light therapy (e.g. pain pump, lap band, penile inflation device, ventriculo-peritoneal shunts, etc.)
  * Known photosensitivity disorder
  * Current active cancer or within one year of cancer treatment or remission
  * Excessive alcohol consumption defined as 14 or more alcoholic drinks per week
  * Serious mental health illness that in the opinion of the investigator would preclude the subject from study participation
  * Active infection, wound or other external trauma to the target area to receive the laser therapy
  * Developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements
  * Participation in a clinical study or other type of research in the past 30 days

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
changes in liver function | 3 months
  measuring liver enzymes (alanine transaminase (ALT) & aspartate aminotransferase (AST) ) and alkaline phosphate before and after low level laser application and the prescribed diet recommendations

SECONDARY OUTCOMES:
changes of lipid profile | 3 months
  measuring effect of low level laser application in addition to diet recommendations on lipid profile (low density lipoprotein LDL, high density lipoprotein HDL, total cholesterol T.C and triglyceride T.G)
changes of Body Mass Index | 3 months
  measuring effect of low level laser application in addition to diet recommendations on body mass index (weight by Kg / height per meter square)
changes of waist circumference | 3 months
  measuring effect of low level laser application in addition to diet recommendations on waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Ebtesam Nabil, doctoral, Principal Investigator — Cairo University
Locations (1):
- Cairo, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol